CLINICAL TRIAL: NCT02803684
Title: Diagnostic Ability of Diffusion MRI and Diffusion Tensor in Renal Graft Biopsies: Pilot Study
Brief Title: Contribution of Diffusion MRI in Renal Graft Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA12065
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Renal Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Whole cohort
  Interventions: Other: MRI examination with tensor diffusion protocol acquisition. No injection needed.

INTERVENTIONS:
Other: MRI examination with tensor diffusion protocol acquisition. No injection needed. — standard MRI examination

SUMMARY:
While renal graft outcomes were really improved for the last decade, long time outcomes remains stable. Indeed, at 10 years after transplantation, the renal graft survival rate reaches 50%. The chronic allograft nephropathy is the main cause of renal graft loss. Other features such as acute allograft rejection, delayed renal recovery and anti-human leukocyte antigen (anti-HLA) antibodies are associated with poor renal graft survival prognosis. Renal graft protocol biopsies at 3 and 12 months after transplantation are valuable to detect precociously renal injuries at a reversible stage before clinical manifestation. However, renal biopsy is an invasive examination with hemorrhagic risk. Diffusion MRI could be a non-invasive diagnostic tool allowing the early detection of renal injuries, especially allograft rejection without hemorrhagic risk. This tool could be applied routinely to the renal allograft recipient in replacement of protocol biopsies.

Here, aim of this study is to correlate the results from diffusion MRI of renal graft with pathologic findings from protocol renal graft biopsies.

In this view, the investigators include prospectively all recipients of renal transplantation who beneficiate of a protocol renal graft biopsy without barrier to peform MRI examination. Thus, the investigators exclude patients who are not be able to beneficiate of a MRI examination and patient obstacle to renal graft biopsy.

Expected results are the Banff classification from the histopathologic analysis of biopsies. The expected results for MRI examination are signal intensity, diffusive coefficient, anisotropy fraction and change of the diffusion way. Next, the investigators search an association between these features by statistical analysis (Wilcoxon test, Chi², Fisher, Pearson or Spearman).

The investigators performed this study since 01/06/2014 and projected end-time to 01/06/2017.

ELIGIBILITY:
Inclusion Criteria:

* Renal graft recipient from Reims hospital
* Over 18 years
* With consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Signal intensity by Diffusion MRI | since transplantation to 12 months after
Banff score (histopathologic findings) | since transplantation to 12 months after

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France